CLINICAL TRIAL: NCT05534308
Title: Effect of Intraoperative Taping on the Control of Edema Resulting From Stripping
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elaine Caldeira de Oliveira Guirro, Clinical professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 12241
Record Dates: First submitted 2022-06-09; First posted 2022-09-09 (Actual); Last update posted 2022-09-09 (Actual); Status verified 2022-09

CONDITIONS: Edema; Varices; Cord
Keywords: Functional Bandages; Edema; Ultrasound; Varices
MeSH Terms: conditions — Edema; Varicose Veins; Cone-Rod Dystrophies

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): The control group (CG) will be composed of patients undergoing the same surgical procedure, and standard treatment consisting only of compression compression by elastic stockings.
  Interventions: Other: No trasoperative taping
- Intervention Group (Experimental): The intervention group (IG) will be composed of patients undergoing phleboextraction with saphenectomy and intervention with contensive taping, in the period intraoperative associated with compression with elastic stockings.
  Interventions: Procedure: Transoperative taping

INTERVENTIONS:
Procedure: Transoperative taping — The intervention group (IG) will be composed of patients undergoing phleboextraction with saphenectomy and intervention with contensive taping, on intraoperative period associated with compression with elastic stockings.
  Arms: Intervention Group
Other: No trasoperative taping — Patients will received only compression stockings after surgery
  Arms: Control Group

SUMMARY:
The aim of the study is to evaluate the effects of the Contensive Taping technique on the control of edema of patients submitted to Phleboextraction Surgery including Saphenectomy.

DETAILED DESCRIPTION:
Edema is a common complication after stripping surgery, so measures that can help the resolution of the condition are important for the recovery in the post operative. The aim of the study is to evaluate the effects of the Contensive Taping technique on the control of edema of patients submitted to phleboextraction surgery including saphenectomy. Therefore, 60 patients of both sexes will be invited to participate in the study, undergoing saphenectomy surgery, divided into two homogeneous groups, determined by the sample calculation. The intervention group (IG) will be composed of patients undergoing phleboextraction with saphenectomy and intervention with contensive taping, in intraoperative period associated with compression with elastic stockings. The control group (CG) will be composed of patients undergoing the same surgical procedure, and standard treatment consisting only of compression by elastic stockings. The procedures for evaluation will be applied before and after seven days of therapeutic intervention. For data analysis, the normality test will be performed and distribution, in addition to a suitable statistical test for the appropriate intra and intergroups, with a significance level of 5%.

ELIGIBILITY:
Inclusion Criteria:

* young adults, aged from 25 to 59 years old, submitted to stripping and saphenectomy.

Exclusion Criteria:

* allergies
* skin lesions
* ulcers.

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-10-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2024-12-20 (Estimated)

PRIMARY OUTCOMES:
Edema | 7 days
  Perimetry (cm)
Dieletric constant | 7 days
  MoistureMeterD

SECONDARY OUTCOMES:
Elasticity | 7 days
  ElastiMeterD
Pain after surgery | 7 days
  Visual Analogue Scale (VAS)
Functionality of Lower Limbs | 7 days
  Lower Extremity Functional Scale (LEFS)
Tissue stiffness | 7 days
  Elastography

CONTACTS AND LOCATIONS:
Overall Officials: Elaine CO Guirro, PhD, Study Director — University of Sao Paulo
Locations (1):
- Medical School of Ribeirão Preto, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No
After the end of Research

REFERENCES:
- [Result] Tatli U, Benlidayi IC, Salimov F, Guzel R. Effectiveness of kinesio taping on postoperative morbidity after impacted mandibular third molar surgery: a prospective, randomized, placebo-controlled clinical study. J Appl Oral Sci. 2020;28:e20200159. doi: 10.1590/1678-7757-2020-0159. Epub 2020 Jul 13. PMID 32667383